CLINICAL TRIAL: NCT07012863
Title: Life-saving Treatment With Dry-plasma for Massive Bleeding in an Pre-hospital Setting - - a Randomized Controlled Study
Brief Title: Life-saving Treatment With Dry-plasma for Massive Bleeding in an Pre-hospital Setting
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBTSB
Record Dates: First submitted 2025-05-26; First posted 2025-06-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-01

CONDITIONS: Bleeding; Aortic Rupture; Gastrointestinal Hemorrhage; Obstetric Bleeding; Blunt Injury; Penetrating Injury
MeSH Terms: conditions — Hemorrhage; Aortic Rupture; Gastrointestinal Hemorrhage; Wounds, Nonpenetrating; Wounds, Penetrating

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients randomized to this arm will get standard treatment within the ambulance service
- Dry plasma (Active Comparator): Patients randomized to this arm will get dry plasma as treatment for the bleeding.
  Interventions: Biological: Dry plasma

INTERVENTIONS:
Biological: Dry plasma — Patient that fulfil the inclusion criteria for this study and are randomized for active treatment will get dry plasma as intervention.
  Arms: Dry plasma

SUMMARY:
The overall goal of this clinical trial is to study how prehospital transfused dry plasma affect outcomes in terms of mortality as well as complications and coagulation status of patients in or about to develop bleeding shock.

Researchers will compare dry plasma to standard care to see if dry plasma improves survival compared to crystalloid fluid in prehospital patients with heavy bleeding.

DETAILED DESCRIPTION:
Major haemorrhage remains one of the leading causes of preventable early death after injury, and the window for effective intervention often closes in the pre-hospital phase. Contemporary European guidelines therefore advocate damage-control resuscitation: permissive hypotension, minimal crystalloid use and early infusion of blood components to avoid dilutional coagulopathy, acidosis and hypothermia. Several reports support that early resuscitation with blood products may save lives.

Freeze- or spray dried plasma containing coagulation factors having up to two years storage time and the possibility of storing ambient temperature, may be an alternative to crystalloids. The results regarding the beneficial results of treatment with plasma are ambiguous. In a previous randomized study using fresh plasma versus crystalloids, 9,8% reduced mortality was shown with resuscitation with plasma. Lower INR and lactate were also seen among the patients treated with plasma. In some studies no effect on mortality could be shown, but in other studies it is suggested that plasma may be beneficial in long transport time.

Acute traumatic coagulopathy can be seen in at least 25 % of severely injured patients who are admitted to a trauma centre. Dilution is often considered as a likely cause although the exact mechanisms and level of aggravation is unknown.

Most studies of prehospital bleeding refer to trauma, but also other causes of bleeding can be severe and even fatal, especially in countries with long distances, e.g. obstetric bleeding, gastrointestinal bleeding and vascular catastrophes.

Hypothesis. The hypothesis of this study is that prehospital treatment with dry plasma to bleeding patients improves the outcome compared to patients receiving standard treatment in terms of lower mortality, lower degree of coagulopathy and less need for blood products when in hospital.

Study aim. The aim of this study is to report outcome for patients receiving standard treatment for major prehospital bleeding compared to patients receiving standard care and to report clinical data for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical signs of bleeding which also triggers resuscitation with crisalloids acording to standard care protocol.

Exclusion Criteria:

* Patients < 18 years of age.
* Patients who lack clinical signs of major bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | Within 24 hours after hospital admission.
  Overall mortality at 24 hours after hospital admission. Will include patients dead at scene or during transportation.

SECONDARY OUTCOMES:
Mortality for patients with bleeding > 500 mL (milliliter) | Within 24 hours after hospital admission
  Specific mortality for patients with a bleeding > 500mL at 24 hours after hospital admission. Will include patients dead at scene or during transport.
Shock Index | baseline, pre-intervention at scene
  Shock Index > 1.3.
Coagulopathy overall | Measured at hospital admission
  PK/INR > 1.2 and/or Platelet count < 150 x 109/L and/or APTT > 34 s or each valuable alone. INR= international normalized ratio PK= prothrombin complex. APTT= activated partial thromboplastin time.

REFERENCES:
- [Derived] Skallsjo G, Wikman A, Wessman C, Sandstrom G. Prehospital Treatment With Dried Plasma in Patients With Major Bleeding-A Prospective Randomised Controlled Multicentre Trial: Statistical Analysis Protocol. Acta Anaesthesiol Scand. 2025 Oct;69(9):e70120. doi: 10.1111/aas.70120. PMID 40910602